CLINICAL TRIAL: NCT07204002
Title: Comparison of Convective Water Vapor Ablation (Convective Water Vapor Energy, WAVE™) With the Rezum™ System Versus Holmium Laser Enucleation of the Prostate (HoLEP) Versus Bipolar Transurethral Resection of the Prostate (TUR-P) in Patients With Benign Prostatic Syndrome (BPS) - A Randomized Study
Acronym: Vektor
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Österreichische Gesellschaft für Urologie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK Nr: 1208/2024
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: BPH (Benign Prostatic Hyperplasia); HoLEP; Rezum; TURP(Transurethral Resection of Prostate)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TURP (Active Comparator)
  Interventions: Procedure: Treatment BPH
- HOLEP (Active Comparator)
  Interventions: Procedure: Treatment BPH
- REZUM (Active Comparator)
  Interventions: Procedure: Treatment BPH

INTERVENTIONS:
Procedure: Treatment BPH — We compare 3 different types of BPH surgery - HoLEP vs. TURP vs. REZUM

SUMMARY:
Benign prostatic enlargement (BPH/BPS) is one of the most common benign diseases in adult men. About 50% of men are affected by the age of 50, and between the ages of 70 and 80 the prevalence rises to 70-80%.

There are various surgical procedures available for the treatment of BPH. In this study, we are investigating three surgical procedures which, based on the current data, appear to be relatively equivalent; however, additional data are still needed to substantiate this.

The aim of this study is to compare the three surgical methods REZUM vs. HoLEP vs. TUR-P for endoscopic transurethral subvesical de-obstruction with regard to both subjective and objective voiding function, as well as improvements in quality of life and sexual function.

The goal of the study is to work out the possible advantages and disadvantages for future patient counseling, thereby defining more precisely the role of these surgical procedures within the armamentarium of urology. This is a single-center, randomized, prospective interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with confirmed benign prostatic syndrome for whom surgical therapy is indicated
* Prostate volume between 30 and 80 ml

Exclusion Criteria:

Lack of capacity to give informed consent

* Emergency surgeries
* Known prostate carcinoma
* Elevated post-void residual urine > 300 ml
* Neurogenic bladder emptying disorder
* Urethral pathologies
* High-intensity anticoagulation
* Dual antiplatelet therapy
* History of pelvic radiation
* Chronic pelvic pain syndrome

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 198 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2030-10-15 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of the surgical techniques in symptom improvement, determined by the change (delta) in the International Prostate Symptom Score (IPSS) at 1 month compared to baseline IPSS. | 1 month